CLINICAL TRIAL: NCT00483301
Title: A Phase II Trial OF Carboplatin, ABI-007 (Abraxane) And Sorafenib (BAY 43-9006) in Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mt. Sinai Medical Center, Miami (Other)
Collaborators: Celgene Corporation (Industry); Bayer (Industry)
Responsible Party: Principal Investigator, Jose Lutzky, Study Principal Investigator, Mt. Sinai Medical Center, Miami
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEL0205
Record Dates: First submitted 2007-05-30; First posted 2007-06-07 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-05

CONDITIONS: Malignant Melanoma
Keywords: Melanoma; Abraxane; Sorafenib; BAY 43-9006; Abraxis
MeSH Terms: conditions — Melanoma | interventions — Sorafenib; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Sorafenib (BAY 43-9006) — dosage
Drug: ABI-007(Abraxane) — dosage

SUMMARY:
The purpose of this study is to compare the effects, good and/or bad, of Carboplatin and ABI-007 (Abraxane) in combination with Sorafenib (BAY 43-9006) on Melanoma.

DETAILED DESCRIPTION:
The primary objective of this phase II multicenter trial is to:

Measure the response rate (RR) of this combination and schedule in patients with metastatic melanoma

The secondary objectives are to:

Assess the safety and toxicity of this regimen in this patient population

Determine the 1-year and median PFS of patients treated according to protocol

Determine overall survival (OS)

STUDY DESIGN

This will be a Phase II study single arm study with a two-stage design with a maximum sample size of 43 patients, 18 in the first stage and 25 in the second stage.

Study duration: A minimum yearly accrual of 10-15 patients/institution is expected. Therefore, to reach the first stage, the study will take 1.2 to 1.8 years with one institution, 0.6 to 0.9 years with 2 institutions, and 0.4 to 0.6 years with 3. If the study continues to full accrual to 43 patients, completion will take 2.9 to 4.3 years with one institution, 1.4 to 2.2 years with two and 0.96 to 1.43 years with three institutions.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of melanoma with measurable disease
* Patients with stage IV, previously untreated, refractory to initial therapy or progressing after response to initial therapy
* Patients with unresectable stage III, including unresectable in-transit metastases
* Two prior chemotherapy regimen is allowed
* One prior immunotherapy regimen is allowed
* No other concurrent investigational therapy
* Radiation therapy to non-target lesions or to one of multiple target lesions may be allowed on a case-by-case basis
* Patients must be past the nadir from previous cytotoxic therapy
* Age at least 18 years
* ECOG performance status 0-2
* Hemoglobin > 9.0 g/dl, absolute neutrophil count (ANC) > 1,500/mm3, platelet count > 100,000/mm3
* Total bilirubin within normal limits, ALT and AST < 2.0 x the ULN ( < 5 x ULN for patients with liver involvement), INR < 1.5 and aPTT within normal limits. Patients who receive anti-coagulation treatment with an agent such as warfarin or heparin may be allowed to participate. For patients on warfarin, close monitoring of at least weekly evaluations will be performed until INR is stable based on a measurement at pre dose, as defined by the local standard of care.
* Creatinine < 1.5 x ULN, serum calcium within normal limits
* Patients with stable brain metastasis who have been treated with either whole brain radiation or Gamma Knife and have been off steroids for > 4 weeks
* Women of childbearing potential and men must agree to use adequate contraception (barrier method of birth control) prior to study entry and for the duration of study participation. Men and women should use adequate birth control for at least three months after the last administration of protocol drugs. Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment.
* Ability to understand and sign a written informed consent document. All patients must have a signed informed consent before registration and initiation of therapy

Exclusion Criteria:

* Cardiac disease: Congestive heart failure > class II NYHA.
* Patients must not have unstable angina (anginal symptoms at rest) or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.
* Uncontrolled hypertension defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management.
* No known severe hypersensitivity or suspected allergy to sorafenib, ABI-007 or any of the excipients
* Patients with neurological symptoms must undergo a CT scan/MRI of the brain to exclude progressing brain metastasis.
* Peripheral neuropathy greater than grade II
* Serious intercurrent medical or psychiatric illness, including serious active infection
* Known human immunodeficiency virus (HIV) infection or chronic Hepatitis B or C.
* Thrombotic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months.
* Pulmonary hemorrhage/bleeding event > CTCAE Grade 2 within 4 weeks of first dose of study drug.
* Any other hemorrhage/bleeding event > CTCAE Grade 3 within 4 weeks of first dose of study drug.
* Serious non-healing wound, ulcer, or bone fracture.
* Evidence or history of bleeding diathesis or coagulopathy
* Major surgery, open biopsy or significant traumatic injury within 4 weeks of first study drug.
* Use of St. John's Wort or rifampin (rifampicin)
* Any condition that impairs patient's ability to swallow whole pills.
* Any malabsorption problem
* No treatment for melanoma within the previous 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2007-05; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Primary Objective | one - two years
  Measure the response rate (RR) of this combination and schedule in patients with metastatic melanoma

SECONDARY OUTCOMES:
Secondary Objective | one-two years
  3.2.1 Assess the safety and toxicity of this regimen in this patient population Determine the 1-year and median PFS of patients treated according to protocol Determine overall survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Lutzky, Physician, Principal Investigator — Mt. Sinai Medical Center Miami Beach Florida
Locations (2):
- United States (2):
  - Dr. Steven O'Day, Los Angeles, California
  - Mt. Sinai Medical Center, Miami Beach, Florida